CLINICAL TRIAL: NCT04911985
Title: Appraisal of the Exactness of a Method to Semiinvasively Evaluate the Cardiac Output of ICU-Patients Through the Use of the Pulsioflex Device
Brief Title: Viability of Pulsioflex Monitoring in ICU
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: proAQT
Record Dates: First submitted 2018-09-17; First posted 2021-06-03 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Cardiogenic Shock
Keywords: Cardiac Output; Cardiac Index; Pulmonary Artery Catheter
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- ICU Patients with PAC: All patients admitted to the Medical ICU of the University Hospital Zürich, complying with the inclusion criteria and monitored by a pilmonary artery catheter
  Interventions: Device: Measurement of the Cardiac Output/ Cardiac Index

INTERVENTIONS:
Device: Measurement of the Cardiac Output/ Cardiac Index — Semiinvasive Measurement of the Cardiac Output/ Cardiac Index with the Pulsion device

SUMMARY:
Goal of the Study is to Study the precision of semi-invasive cardiac index monitoring by means of the ProAQT (PULSION Medical Systems SE) sensor, whereby the pulmonary artery catheter will serve as gold standard.

DETAILED DESCRIPTION:
Goal of the Study is to Study the precision of semi-invasive cardiac index monitoring by means of the ProAQT (PULSION Medical Systems SE) sensor, whereby the pulmonary artery catheter will serve as gold standard.

Measurements will be performed contemporaly with both devices every 4 hours and all clinical and hemodynmaic parameters will be recorded, including but not limited to central venous pressure, wege pressure, mechanical ventilation pressures, blood pressures, volume balance as well as vasoaktive medikation doses. This precise evaluation shall serve to evaluate the precision of the ProAQT to estimate the cardiac index under different clinical situation in the intensive care unit. A precision difference of below 30% between both methods will be regarded as clinically irrelevant, suggesting equipoise between both methods.

ELIGIBILITY:
Inclusion Criteria:

* In situ pulmonary artery catheter
* Above 16 years of age
* At least 36 hours of continuous hemodynamic monitoring with the pulmonary artery catheter planed

Exclusion Criteria:

* Patients with:
* Permanent or pesisting Atrial Fibrilation or Ventricular Arrythmias
* Moderate to Severe Aortic Insuficiency or Aortic Stenosis
* Intravascular Cardiac Assist Device
* Planed removal of the pulmonary artery catheter <36 hours

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients admitted to the Medical ICU of the University Hospital Zürich complying with the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Bias of proAQT measurement | 51 Hours
  Bias between the Pulsion CI measurement and the gold standard CI measurement by Pulmonary artery catheterisation

SECONDARY OUTCOMES:
Percentage Error of CI Measurement | 51 Hours
  Percentage Error of CI Measurement between Pulsion and PAC measurement

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Medical intensive care unit, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ameloot K, Van De Vijver K, Broch O, Van Regenmortel N, De Laet I, Schoonheydt K, Dits H, Bein B, Malbrain ML. Nexfin noninvasive continuous hemodynamic monitoring: validation against continuous pulse contour and intermittent transpulmonary thermodilution derived cardiac output in critically ill patients. ScientificWorldJournal. 2013 Nov 11;2013:519080. doi: 10.1155/2013/519080. eCollection 2013. PMID 24319373
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Bland JM, Altman DG. Measuring agreement in method comparison studies. Stat Methods Med Res. 1999 Jun;8(2):135-60. doi: 10.1177/096228029900800204. PMID 10501650
- [Background] Broch O, Carbonell J, Ferrando C, Metzner M, Carstens A, Albrecht M, Gruenewald M, Hocker J, Soro M, Steinfath M, Renner J, Bein B. Accuracy of an autocalibrated pulse contour analysis in cardiac surgery patients: a bi-center clinical trial. BMC Anesthesiol. 2015 Nov 26;15:171. doi: 10.1186/s12871-015-0153-2. PMID 26612072
- [Background] Smetkin AA, Hussain A, Kuzkov VV, Bjertnaes LJ, Kirov MY. Validation of cardiac output monitoring based on uncalibrated pulse contour analysis vs transpulmonary thermodilution during off-pump coronary artery bypass grafting. Br J Anaesth. 2014 Jun;112(6):1024-31. doi: 10.1093/bja/aet489. Epub 2014 Feb 13. PMID 24531685